CLINICAL TRIAL: NCT05932342
Title: Improving Cognition of Older Adults in Community Housing (I-COACH)
Brief Title: Improving Cognition of Older Adults in Community Housing
Acronym: I-COACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: LOFT Community Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 027 - 2023
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-09

CONDITIONS: Aging; Mental Disorder
Keywords: cognitive remediation; social activity; exercise; aging; community
MeSH Terms: conditions — Mental Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention will be provided over 3 iterative group of 6 participants each
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Integrated program of cognitive remediation, physical exercise and socially- stimulating activity (Experimental): Cognitive Remediation (CR) is a well-established intervention that aims to improve neurocognitive abilities (such as memory performance, executive functioning, processing speed, and attention) using four techniques: didactic teaching, computerized drills, in-class strategic monitoring and discussions of the generalization of cognitive skills to daily life.
  The physical exercise component consists of physical activities designed for the geriatric population that aim to reduce sedentary behaviors while increasing social engagement.
  The socially stimulating activity aim to decrease social isolation, improve well-being, community connection and rapport.
  The integrated, 12-week, group-based program consists of CR 1h/day, 2 days/week, 30min of physical exercises 1day/week and 1h of socially stimulating activities 1day/week
  Interventions: Behavioral: Integrated program of cognitive remediation, physical exercise and socially stimulating activity

INTERVENTIONS:
Behavioral: Integrated program of cognitive remediation, physical exercise and socially stimulating activity — Cognitive Remediation (CR) is a well-established intervention that aims to improve neurocognitive abilities (such as memory performance, executive functioning, processing speed, and attention) using four techniques: didactic teaching, computerized drills, in-class strategic monitoring and discussions of the generalization of cognitive skills to daily life.
  The physical exercise component consists of physical activities designed for the geriatric population that aim to reduce sedentary behaviors while increasing social engagement.
  The socially stimulating activity aim to decrease social isolation, improve well-being, community connection and rapport.

SUMMARY:
The I-COACH study will focus on seniors with mental health conditions who are living in senior community housing. This initiative proposes to assess the feasibility and acceptability of a 12-week integrated program of cognitive remediation (CR) in combination with social and physical activity using an open-label design. The program will be provided over three iterative groups of six participants each, with one Personal Support Worker (PSW). The program will be co-designed at a granular level in an iterative process, drawing upon feedback provided by each participant group, PSW, and community housing staff to improve the user experience.

We will build the capacity for community personal support workers (PSWs) to deliver this program independently and with fidelity to the intervention model. Our ultimate goal is to help seniors continue to live as long as possible in their homes within the community.

DETAILED DESCRIPTION:
This project entails the development and implementation of a12-week integrated program of cognitive remediation (CR) in combination with social and physical activity of 18 older adults living in senior housing.

The study will be recruiting individuals, age 50 or older, who meet criteria for any Diagnostic and Statistical Manual of Mental Disorders (DSM)-V diagnosis and are living in community housing.

Participants will be recruited from five senior housing units. Prior to enrollment, participants will undergo a baseline assessment consistent of neuropsychological assessment (NP). Once enrolled, each participant will participate in the 12 - weeks program. The program will be offered 4 days per week and will consist of 2 days of 1-hour CR training, one day of 30 min physical activity and one day of 1-hour social activity. The intervention will be delivered by the research team and the senior community housing PSWs. The PSWs involved in the study are part of the participant's circle of care and will be trained and operating under supervision in collaboration with the research team.

Following the completion of the 12-week program, group participants and staff will be invited to complete a satisfaction survey and the System Usability Scale (SUS) to gauge their feedback to the program and also to complete a semi-structured interview involving a qualitative assessment.

Primary Aim:

To design a feasible and tolerable active program for seniors living in the community setting.

Secondary Aim:

To modify CR using an iterative process that meets the capacity of senior community housing PSWs to deliver CR independently.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years and above. The rationale of age cutoff of 50 is that this age is considered a typical geriatric age cutoff especially for people with severe mental illness
2. Any race or ethnicity
3. Any gender identity
4. Meets DSM-V criteria for any disorder
5. Clinically stable as operationalized by (1) having not been admitted to a psychiatric hospital within the 3 months prior to assessment, (2) having had no change in psychotropic medication dosage within the 4 weeks prior to assessment, and (3) ascertained to be clinically and medically stable by one the study psychiatrists.
6. Willingness and ability to speak English
7. Willingness to provide informed consent or assent as applicable.
8. Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice. Both vision and hearing ability will be assessed by asking the participant if they can see the text and hear the research personnel during the screening consent and enrolment process.

Exclusion Criteria:

1. Meets diagnostic criteria for active substance use or dependence within the 6 months prior to the initial assessment except for caffeine or nicotine
2. Has profound cognitive impairment that, in the opinion of the PI, precludes benefit from CR and therefore study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Participant's satisfaction | end of week 12 of the intervention
  This is measured using the Satisfaction Survey which assesses participants' agreement on 10 statements each measuring the degree of agreement or disagreement of participants using a 7-point Likert Scale. Minimum score is 10 and maximum score is 70. Higher scores indicate better satisfaction.
Acceptability and Usability of Cognitive Remediation | end of week 12 of the intervention
  This is assessed using the System Usability Scale (SUS). The scale is comprised of 10 statements each measuring the degree of agreement or disagreement of participants using 5 -point Likert Scale. Minimum score is 0 and maximum is 100. Higher scores indicate better usability.
Participants' feedback of the program | end of week 12 of the intervention
  Semi-structured qualitative interview
Staff Feedback of the program | Within one week from the end of week 12 of the intervention
  Semi-structured qualitative interview
Sessions and overall program attendance | end of week 12 of the intervention
  Attendance logs

SECONDARY OUTCOMES:
Staff Feedback of the delivery of the program | Within one week from the end of week 12 of the intervention
  Semi-structured qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Angela Golas, MD, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilmer T, Ojeda VD, Folsom D, Fuentes D, Criado V, Garcia P, Jeste DV. Costs of community-based public mental health services for older adults: variations related to age and diagnosis. Int J Geriatr Psychiatry. 2006 Dec;21(12):1121-6. doi: 10.1002/gps.1616. PMID 16977681
- [Background] Bangor A, Kortum PT,Miller JT: An Empirical Evaluation of the System Usability Scale. International Journal of Human Computer Interaction 2008; 24:574-594
- [Background] Arrieta H, Rezola-Pardo C, Echeverria I, Iturburu M, Gil SM, Yanguas JJ, Irazusta J, Rodriguez-Larrad A. Physical activity and fitness are associated with verbal memory, quality of life and depression among nursing home residents: preliminary data of a randomized controlled trial. BMC Geriatr. 2018 Mar 27;18(1):80. doi: 10.1186/s12877-018-0770-y. PMID 29580209
- [Background] Gremeaux V, Gayda M, Lepers R, Sosner P, Juneau M, Nigam A. Exercise and longevity. Maturitas. 2012 Dec;73(4):312-7. doi: 10.1016/j.maturitas.2012.09.012. Epub 2012 Oct 11. PMID 23063021
- [Background] Vagetti GC, Barbosa Filho VC, Moreira NB, Oliveira Vd, Mazzardo O, Campos Wd. Association between physical activity and quality of life in the elderly: a systematic review, 2000-2012. Braz J Psychiatry. 2014 Jan-Mar;36(1):76-88. doi: 10.1590/1516-4446-2012-0895. Epub 2014 Jan 17. PMID 24554274
- [Background] Glass TA, De Leon CF, Bassuk SS, Berkman LF. Social engagement and depressive symptoms in late life: longitudinal findings. J Aging Health. 2006 Aug;18(4):604-28. doi: 10.1177/0898264306291017. PMID 16835392
- [Background] Cornwell EY, Waite LJ. Social disconnectedness, perceived isolation, and health among older adults. J Health Soc Behav. 2009 Mar;50(1):31-48. doi: 10.1177/002214650905000103. PMID 19413133
- [Background] McHugh JE, Lawlor BA. Exercise and social support are associated with psychological distress outcomes in a population of community-dwelling older adults. J Health Psychol. 2012 Sep;17(6):833-44. doi: 10.1177/1359105311423861. Epub 2011 Nov 22. PMID 22108290
- [Background] Krivanek TJ, Gale SA, McFeeley BM, Nicastri CM, Daffner KR. Promoting Successful Cognitive Aging: A Ten-Year Update. J Alzheimers Dis. 2021;81(3):871-920. doi: 10.3233/JAD-201462. PMID 33935078
- [Background] Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. Ageing Res Rev. 2013 Jan;12(1):263-75. doi: 10.1016/j.arr.2012.07.003. Epub 2012 Jul 25. PMID 22841936
- [Background] Golas AC, Kalache SM, Tsoutsoulas C, Mulsant BH, Bowie CR, Rajji TK. Cognitive remediation for older community-dwelling individuals with schizophrenia: a pilot and feasibility study. Int J Geriatr Psychiatry. 2015 Nov;30(11):1129-34. doi: 10.1002/gps.4329. Epub 2015 Aug 6. PMID 26250542
- [Background] Harvey PD, Bowie CR. Cognitive enhancement in schizophrenia: pharmacological and cognitive remediation approaches. Psychiatr Clin North Am. 2012 Sep;35(3):683-98. doi: 10.1016/j.psc.2012.06.008. Epub 2012 Jul 15. PMID 22929873
- [Background] Kurtz MM. Cognitive remediation for schizophrenia: current status, biological correlates and predictors of response. Expert Rev Neurother. 2012 Jul;12(7):813-21. doi: 10.1586/ern.12.71. PMID 22853789
- [Background] HAPPYneuron I: Scientific Brain Training PRO, Campbell, CA, USA, 2009.